CLINICAL TRIAL: NCT06305247
Title: An Open-label, Phase I/IIa First-in-human, Dose Escalation and Cohort Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetic, Pharmacodynamic and Antitumour Activity of ERK1/2 Inhibitor IPN01194 as Single Agent in Adult Participants With Advanced Solid Tumours
Brief Title: A Study to Assess IPN01194 When Administered Alone in Adults With Advanced Solid Tumours
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CLIN-01194-450; 2023-506228-10-00 (Other: Ipsen)
Record Dates: First submitted 2024-02-27; First posted 2024-03-12 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Melanoma; Head and Neck Squamous Cell Carcinoma; Pancreatic Ductal Adenocarcinoma; Colorectal Cancer; Solid Tumor
MeSH Terms: conditions — Melanoma; Squamous Cell Carcinoma of Head and Neck; Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Phase I is a dose escalation with backfill in participants with selected MAPKm advanced solid tumours.
  Phase IIa (cohort expansion) is an open label randomised study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase I (Dose Escalation with Backfilling) (Experimental): Nine dose levels are planned to be tested.
  Interventions: Drug: IPN01194
- Phase IIa (Cohort Expansion) (Experimental): Study intervention will be administered at one of two doses of interest determined at the end of Phase I.
  Interventions: Drug: IPN01194

INTERVENTIONS:
Drug: IPN01194 — IPN01194 will be taken orally over a period of 28 days (a "Cycle") at the assigned dose level. The dose limiting toxicity (DLT) observation period consists of the first 28 days of treatment with IPN01194 (Cycle 1).
  Participants will receive IPN01194 treatment beyond Cycle 1 until treatment is precluded by toxicity, disease progression, or upon participant's request or investigator decision.
  Arms: Phase I (Dose Escalation with Backfilling)
Drug: IPN01194 — All participants will receive IPN01194 orally for 28-day cycles at one of the two dose levels determined at the end of Phase I.
  Participants will receive IPN01194 treatment until treatment is precluded by toxicity, disease progression, or upon participant's request or investigator decision
  Arms: Phase IIa (Cohort Expansion)

SUMMARY:
The purpose of this study is to determine the appropriate dosage, safety and effectiveness of the study drug, IPN01194 in adults with advanced solid tumours.

The participants in this study will have advanced solid tumours. 'Advanced solid tumours' refers to cancers that can occur in several places, including cancers in organs or tissues that have spread from their original site to nearby tissues or other parts of the body.

In this study, all participants will receive the study drug, which will be taken by mouth (orally).

DETAILED DESCRIPTION:
The study consists of two parts, called Phase I and Phase IIa.

Phase I is designed to assess the safety of increasing doses of IPN01194 in participants with specific types of advanced solid tumours.

The aim of this "dose escalation" phase is to find the dose range showing activity on the tumor that can be tolerated by the participants, and to determine the two doses for further testing in Phase IIa. Phase I will assess how the body processes and responds to the study drug when administered with and without food.

In Phase IIa, participants with selected single tumour type will be invited to take part. During this phase, the two dose levels of the study drug identified from Phase I will be tested. Participants will take the study drug one of the two dose levels. Each participant will be assigned to a dose level at random (by chance).

Each phase will consist of three periods:

1. A period to assess eligibility (screening period) that will take up to 28 days.
2. A treatment period of at least 28 days that will require at least two visits for the first month followed by one visit every month. There will be also one visit, at the end of treatment, at least 30 days after the last administration of study drug.
3. A follow-up period (Phase IIa participants only), where every 3 months, participants will be contacted by phone, until death or the study cut-off date, whichever comes first.

Participants will undergo blood samplings, urine collections, physical examinations, and clinical evaluations. They may continue some other medications, but the details need to be recorded.

If in the opinion of the investigator a participant is continuing to experience clinical benefit after the cut-off date, the participant may remain in the study and continue to receive the study drug until either disease progression, unacceptable toxicity or other withdrawal criteria are met.

ELIGIBILITY:
Inclusion Criteria :

* Participants must be ≥18 years of age
* Participants with histologically confirmed metastatic solid tumour (melanoma, metastatic colorectal cancer (CRC), pancreatic ductal adenocarcinoma (PDAC) or head and neck squamous cell carcinoma (HNSCC)) for whom no suitable alternative standard therapy exists.
* Participants must bear tumours harbouring selected classes of genetic mutations, (MAPKm).
* Participants must have measurable disease per Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1
* Eastern Cooperative Oncology Group (ECOG)/performance status (PS) of 0 or 1.
* Participants must consent to the use of archival tumour tissue or, if not available, collection of fresh tumour biopsy at screening
* Male and female participants Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical trials.

Exclusion Criteria

* Gastrointestinal conditions that could impair absorption of IPN01194 or inability to swallow oral medications.
* Any evidence of severe active infection or inflammatory condition.
* Non-adequate cardiac function
* Have one or more of study defined ophthalmological findings/conditions
* Known psychiatric or substance abuse disorder, or any other cognitive disorder per the opinion of the investigator that would interfere with the participant's ability to cooperate with the requirements of the study.
* Underlying medical conditions that, in the investigator's or sponsor's opinion, will obscure the interpretation of toxicity determination or AEs.
* Known second malignancy within the last 2 years prior to first dose of study intervention..
* Major surgery within 28 days prior to first dose of study intervention.
* Ongoing AEs caused by any prior anti-cancer therapy ≥Grade 2 (National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0).
* Active brain metastases or leptomeningeal metastases
* Current enrolment or past participation in any other clinical trial involving an investigational study treatment within the last 28 days.
* Live vaccine(s) within 28 days prior to first dose of study intervention
* Concurrent treatment with any other anti-cancer therapy (including radiotherapy or investigational agents).
* Treatment with medications that prolong the QT/QTc interval.
* Treatment with strong and moderate CYP3A4 inducers
* Treatment with strong or moderate inhibitors of CYP3A4
* Only for Phase I participants assigned to dose escalation and low-dose backfill participants: treatment with proton pump inhibitors within 14 days prior to first dose of study intervention.
* Non-adequate bone marrow function
* Non-adequate renal function
* Non-adequate hepatic function
* Non adequate coagulation function.
* Known uncontrolled human immunodeficiency virus (HIV) infection or hepatitis B or C
* Sensitivity to IPN01194 or any of its components.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-04-03 (Actual); Primary Completion 2028-03-20 (Estimated); Study Completion 2028-03-20 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Percentage of participants with dose limiting toxicity (DLT) | Within 28 days of first dose
Phase 1: Percentage of participants experiencing Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TE SAEs) | At 30 days following the last administration of study intervention
  An Adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Phase 1: Percentage of participants with dose interruptions and permanent treatment discontinuations | At 30 days following the last administration of study intervention
Phase 2a: Objective response rate (ORR) | At end of treatment (up to approximately 32 months)
  Defined as the percentage of participants with best overall response (BOR) of complete response (CR) or partial response (PR) as determined by investigator.

SECONDARY OUTCOMES:
Phase 1: Time to maximum observed drug concentration (Tmax) after single and multiple doses of IPN01194 | At Day 1 and Day 15.
Phase 1: Maximum observed drug concentration (Cmax) after single and multiple doses of IPN01194 | At Day 1 and Day 15.
Phase 1: Area under the plasma concentration time curve (AUCtau) after single and multiple doses of IPN01194 | At Day 1 and Day 15.
  AUCtau is defined as the concentration of drug over one dosing interval.
Phase 1: Geometric mean ratio of Cmax of IPN01194 administered in fed state relative to fasted state | Between Day -8 and Day -3 (fasted period) and between Day -10 and Day -7 (fed state period)
Phase 1: Geometric mean ratio of AUClast of IPN01194 administered in fed state relative to fasted state | Between Day -8 and Day -3 (fasted period) and between Day -10 and Day -7 (fed state period)
  AUClast is defined as the concentration of drug from time zero to the last observable concentration.
Phase 1: Geometric mean ratio of AUCinf administered in fed state relative to fasted state | Between Day -8 and Day -3 (fasted period) and between Day -10 and Day -7 (fed state period)
  AUCinf is defined as the concentration of drug extrapolated to infinite time.
Phase 1: Prolongation of corrected QT interval (QTc) | Within 28 days of first dose
  Prolongation of QTc defined as the upper limit of 90% confidence interval for change from baseline QTc evaluated over Cycle 1 at the highest clinically relevant exposure.
Phase 1: Objective response rate (ORR) | At end of treatment (up to approximately 32 months)
  The ORR is defined as the percentage of participants with best overall response (BOR) of complete response (CR) or partial response (PR).
Phase 2a: Duration of response (DoR) | From randomisation to end of treatment (up to approximately 32 months)
  Defined as the percentage of participants with BOR of CR or PR, as determined by investigator per RECIST version 1.1
Phase 2a: Progression-free survival (PFS) | From randomisation to end of treatment (up to approximately 32 months)
  PFS is defined as the time from the date of randomisation to the date of the first documented disease progression, as determined by investigator per RECIST version 1.1.
Phase 2a: PFS rate at 4 months | From randomisation to 4 months
Phase 2a: Disease control rate (DCR) | At end of treatment (up to approximately 32 months)
  DCR is defined as the percentage of participants with BOR of CR, PR or stable disease (SD), as determined by investigator per RECIST version 1.1.
Phase 2a: Percentage of participants with TEAEs and TE SAEs | At end of treatment (up to approximately 32 months)
Phase 2a: Percentage of participants with dose interruptions and permanent treatment discontinuations | At end of treatment (up to approximately 32 months)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (12):
- United States (5):
  - The Angeles Clinic and Research Institute - California, Los Angeles, California
  - UC San Diego Health System - La Jolla, San Diego, California
  - Yale Cancer Center - New Heaven, New Haven, Connecticut
  - Sarah Cannon Research Institute (SCRI) - Nashville, Nashville, Tennessee
  - Virginia Cancer Specialist, Fairfax, Virginia
- France (4):
  - Centre Léon Bérard - Lyon, Lyon
  - Paris Saint-Louis, Paris
  - Institut de Cancerologie de l'Ouest (St-Herblain), Saint-Herblain
  - IGR-Villejuif, Villejuif
- Spain (3):
  - Barcelona - Val D'Hebron, Barcelona
  - Fundacion Jimenez Diaz - Madrid, Madrid
  - M.D. Anderson Cancer Center Madrid, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications.
  Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and/or EU.
Access Criteria: Further details on Ipsen's sharing criteria and process for sharing are available here (https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/).
URL: https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/